CLINICAL TRIAL: NCT04611308
Title: The Role of C1q Tumor Necrosis Factor-related Protein 6 (CTRP6) in Breast Cancer
Brief Title: The Role of C1q Tumor Necrosis Factor-related Protein 6 in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samia Farouk Hamed Ahmed, Samia Farouk Hamed Ahmed, Assiut University
Other Study IDs: CTRP6 in Breast Cancer
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases
  Interventions: Other: C1q tumor necrosis factor-related protein 6 levels
- controls
  Interventions: Other: C1q tumor necrosis factor-related protein 6 levels

INTERVENTIONS:
Other: C1q tumor necrosis factor-related protein 6 levels — C1q tumor necrosis factor-related protein 6 is a tumor marker

SUMMARY:
Globally, breast cancer is one of the most prevalent cancers in women and is the second leading cause of cancer death , representing 15% of worldwide deaths per year . In Egypt, it accounts for 32 % of cancer in women with a high mortality rate.

DETAILED DESCRIPTION:
Globally, breast cancer is one of the most prevalent cancers in women and is the second leading cause of cancer death , representing 15% of worldwide deaths per year. In Egypt, it accounts for 32 % of cancer in women with a high mortality rate.

The etiology of breast cancer is multifactorial in which multiple epigenetic and genetic variations affect its incidence and prognosis . Although diagnostic methods and therapeutic strategies for breast cancer have been improved in past decades, long-term survival of breast cancer patients still remains poor due to high proliferation, metastasis and post-surgical recurrence rate.

Therefore, it is critical to develop more effective screening methods that can detect BC at an early stage and novel therapeutic targets for better treatment. This may be achieved by understanding the molecular mechanisms underlying the initiation and progression of this malignancy.

Complement C1q tumor necrosis factor-related protein (CTRPs) are a protein family of adiponectin paralogs which contains fifteen members, CTRP1- CTRP15. This super family are involved in several biological processes, including metabolism, immunity, inflammation, apoptosis and cell differentiation (15, 16). Accumulating evidence correlates CTRP family members with carcinogenesis and signaling pathways associated with cancer development, progression and metastasis.

C1q tumor necrosis factor-related protein 6 (CTRP6) or (C1qTNF6) is a member of CTRPs family. It contains four domains including signal peptide, short N-terminal variable region, collagen domain and C-terminal C1q domain. It is expressed mainly in placenta, heart, uterus and adipose tissue.

CTRP6 is involved in multiple physiological processes, such as regulating cell proliferation and differentiation. It also mediates fatty acid oxidation, adipogenesis and insulin sensitivity, attenuates cell fibrosis and displays anti-inflammatory properties.

Although recent studies have revealed that adiponectin has an inhibitory role in carcinogenesis, the role of CTRP6 in carcinogenesis remains unclear. CTRP6 was initially found to be overexpressed and possibly contributes to tumor angiogenesis in many hepatocellular carcinomas. Moreover, recent research indicates that CTRP6 is correlated with gastric cancer progression by mediating proliferation, migration and apoptosis, which reveals a similar pattern in lung adenocarcinoma.

However, tumor suppressor functions of CTRP6 were also successively reported. CTRP6 was found to have inhibitory effect on the proliferation and migration of ovarian cancer cells. Moreover, CTRP6 significantly suppressed the growth and invasion activity of the oral squamous cell carcinoma cells.

The role CTRP6 plays in breast cancer is yet unknown. The present study will investigate the level of CTRP6 in BC specimens. Furthermore, the pathological functions of CTRP6 in BC, including cell growth, proliferation, migration, and effect on inflammation and angiogenesis will be studied in breast cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older.
* Newly diagnosed patients with histopathological confirmation of the diagnosis of breast cancer at any stage.

Exclusion Criteria:

* Patients with a prior history of other cancers.
* Patients with more than one cancer.
* Patients treated with chemotherapy or radiotherapy before initial samples collection.
* Pregnant women.
* Patients with unqualified or insufficient data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Approximately 102 cases.
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the CTRP6 levels in breast cancer. | 1 October 2021